CLINICAL TRIAL: NCT04362267
Title: Incidence of SARS-Cov2 Infection Among HCW in Lille University Hospital
Brief Title: Longitudinal Study of Covid-19 Infection Among HCW in a French University Hospital
Acronym: PRECOVIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Fondation Santé Roquette (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020_34; 2020-A00950-39 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-04

CONDITIONS: Sars-CoV2
Keywords: Incidence; Health Care Workers; occupational exposure; environmental exposure; serological testing; RT-PCR
MeSH Terms: interventions — COVID-19 Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: self-administered questionnaire — Every14 days, clinical and occupational questionnaire are performed among a cohort of HCW exposed to covid occupational exposure
  Other Names: a specifically designed self-administered questionnaire
Diagnostic Test: SARS-Cov2 testing — Every14 days, SARS-Cov2 RT-PCR, serological testing are performed among a cohort of HCW exposed to covid occupational exposure

SUMMARY:
The aim of the study is to determine the incidence o of SARS-cov2 infection among health care workers highly exposed to covid 19 during 10 weeks et to analyze the determinants of their occupational and environmental exposure. Every 14 days, we performed SARS-Cov2 RT- PCR, serological testing and clinical questionnaire among a cohort of 100 HCW with a high degree of exposure to covid19 infection. Information about occupational exposure as the workplace, the activity of care, the characteristics of patient infected are captured, as well as environmental or personal exposure.

The results will support the design of a new care organization and will define new ways of protection for patients (covid or not covid 19) and prevention for HCW.

ELIGIBILITY:
Inclusion Criteria:

- Health Care workers with covid high exposure during the care activities

Exclusion Criteria:

* Heath Care Worker with SARS-Cov2 infection ( RT-PCR +) or SARS-Cov2 immunity in serological testing
* HCW off work
* Subjects on leave

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Care workers exposed to covid occupational exposure
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
the incidence of SARS- Cov2 infection Heath Care Worker diagnosed by the positivity of SARS-Cov2 RT-PCT and serological testing | at 14 weeks

SECONDARY OUTCOMES:
the incidence of SARS- Cov2 infection Heath Care Worker diagnosed by the positivity of SARS-Cov2 RT-PCT and serological testing | once every 14 days for an average of 14 weeks
Occupational exposures associated with the SARS-Cov2 infection | once every 14 days for an average of 14 weeks
Environmental exposures associated with the SARS-Cov2 infection | once every 14 days for an average of 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Annie SOBASZEK, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France